CLINICAL TRIAL: NCT05946486
Title: Phase III Randomized, Multicenter Open Label Study to Evaluate the Efficacy of Immunomodulatory Therapy in Case of Psychiatric Disorders With Proven Dysimmunity.
Brief Title: Evaluation of the Efficacy of Immunomodulatory Therapy in Case of Psychiatric Disorders With Proven Dysimmunity.
Acronym: TIM-DePisT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2019/59
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Mental Disorder
Keywords: psychotic disorders; pathogenic central nervous system (CNS) autoantibodies; immunomodulatory therapy
MeSH Terms: conditions — Mental Disorders; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): continuation of ongoing psychiatric care (with or without standard treatment as usual (i.e. antipsychotics, mood stabilisers, antidepressants and/or anxiolytics)).
- experimental group (Experimental): immunomodulatory treatment by rituximab, 1g for adults or 375 mg/m2 for children, renewed at 14 days (+/- 3 days), added to stable ongoing psychiatric care (with or without standard treatment as usual ( i.e. antipsychotic, mood stabiliser, antidepressant and/or anxiolytic)). The rituximab is the best immunomodulatory treatment recommended for neurologic encephalitis.
  Interventions: Drug: immunomodulatory treatment by rituximab

INTERVENTIONS:
Drug: immunomodulatory treatment by rituximab — 1g for adults or 375 mg/m2 for children, renewed at 14 days (+/- 3 days)
  Arms: experimental group

SUMMARY:
This is an open phase III randomized clinical trial studying the superiority of management by immunomodulator treatment of psychiatric disorders (psychosis and bipolar disorders) for patients previously identified as carriers of autoimmunity such as as the presence of a pathogenic anti-glutamatergic NMDA receptor antibody (NMDAr-Ac).

DETAILED DESCRIPTION:
This is an open phase III randomized clinical trial studying the superiority of management by immunomodulator treatment of psychiatric disorders (psychosis and bipolar disorders) for patients previously identified as carriers of autoimmunity such as as the presence of a pathogenic anti-glutamatergic NMDA receptor antibody (NMDAr-Ac). The aim is to assess the clinical efficacy of this treatment associated with the usual recommended psychotropic treatment. To meet this objective, we will use, via a National Center for Scientific Research (CNRS) Research laboratory in Bordeaux, a very sensitive diagnostic platform to detect and demonstrate the pathogenesis of antibodies in patient serum. This platform is operational only within the framework of validation of the results by the reference center for neurological autoimmune diseases in Lyon

ELIGIBILITY:
Inclusion Criteria:

* For Adult: First acute or relapse of psychotic disorders defined by the BPRS-E scale with or without standard pharmacological treatment.
* For Children: Child over 6 years old with a first acute or relapse of psychotic disorders defined by the Kiddie sads-PL scale with or without standard pharmacological treatment.
* Biological diagnosis of pathogenic CNS autoantibodies in the blood.
* MDC scale score >3 is required for inclusion in step 2.
* Normal ECG in case of previous heart disease.
* Informed consent of the patient or his legal representatives.
* Effective contraception for women of childbearing potential during the study and for at least 12 months after the last rituximab administration.

Exclusion Criteria:

* Developmental disorder related to a genetic disease.
* Co-existing disorder of severe neurological disease.
* Chronic psychotic disorders receiving ongoing neuroleptic treatment with efficacy.
* Hypersensitivity to the active substance (rituximab) or to murine proteins, or to any of the other excipients
* Blood platelets < 75x109/L
* Neutrophils < 1.5x109/L
* Neoplastic pathology,
* Hepatitis B or HIV infection,
* Contraindication to immunosuppressant treatment (active severe infection, severely immunocompromised state).
* Severe heart failure (New York Heart Association Class IV) or severe, uncontrolled cardiac disease
* Pregnant or breastfeeding women
* Currently receiving an investigational drug or received an investigational drug or device within 30 days (or 5 half-lives for drugs, whichever is longer) prior to screening.
* Previous treatment with rituximab in the past 12 months.
* Patients with a history of recurring or chronic infections or with underlying conditions which may further predispose them to serious infection (e.g. hypogammaglobulinemia).
* Recent vaccination with live viral vaccine (within 3 months).
* Any other medical illness or disability that, in the opinion of the investigator, would compromise effective trial participation.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Adult patients : the remission of psychiatric symptoms at 3 months | 3 months after randomization
  The primary endpoint outcome is the remission of psychiatric symptoms at 3 months, defined as:
  - For adult patients: 20% decrease from baseline of Brief psychiatric rating scale-Extended (BPRS-E scale).
Minor patients : the remission of psychiatric symptoms at 3 months | 3 months after randomization
  The primary endpoint outcome is the remission of psychiatric symptoms at 3 months, defined as:
  - For patients <18years or adults patients included at adolescent age at 2nd step inclusion visit: clinically significant difference ≤3 from baseline of CBCL/6-18 (Child Behavior Checklist) scale.

SECONDARY OUTCOMES:
Adult Patients : the remission of psychiatric symptoms at 12 months | 12 months after randomization
  the remission of psychiatric symptoms defined as:
  - For adult patients: 20% decrease from baseline of Brief psychiatric rating scale-Extended (BPRS-E scale).
Adult Patients : the remission of psychiatric symptoms at 6 months | 6 months after randomization
  the remission of psychiatric symptoms defined as:
  - For adult patients: 20% decrease from baseline of Brief psychiatric rating scale-Extended (BPRS-E scale).
Adult Patients : the remission of psychiatric symptoms at 1 month | 1 month after randomization
  the remission of psychiatric symptoms defined as:
  - For adult patients: 20% decrease from baseline of Brief psychiatric rating scale-Extended (BPRS-E scale).
Minor patients : the remission of psychiatric symptoms at 12 months | 12 months after randomization
  The primary endpoint outcome is the remission of psychiatric symptoms at 12 months, defined as:
  - For patients <18years or adults patients included at adolescent age at 2nd step inclusion visit: clinically significant difference ≤3 from baseline of CBCL/6-18 (Child Behavior Checklist) scale.
Minor patients : the remission of psychiatric symptoms at 6 months | 6 months after randomization
  The primary endpoint outcome is the remission of psychiatric symptoms, defined as:
  - For patients <18years or adults patients included at adolescent age at 2nd step inclusion visit: clinically significant difference ≤3 from baseline of CBCL/6-18 (Child Behavior Checklist) scale.
Minor patients : the remission of psychiatric symptoms at 1 month | 1 month after randomization
  The primary endpoint outcome is the remission of psychiatric symptoms, defined as:
  - For patients <18years or adults patients included at adolescent age at 2nd step inclusion visit: clinically significant difference ≤3 from baseline of CBCL/6-18 (Child Behavior Checklist) scale.
Adult patients : general functioning at 1 month | 1 month after randomization
  for Global assessment of functioning scale (GAF scale), a mean score of 60 and above is expected to be achieved indicating patients experiencing mild to moderate symptoms and functioning pretty well in daily life.
Adult patients : general functioning at 3 months | 3 months after randomization
  for Global assessment of functioning scale (GAF scale), a mean score of 60 and above is expected to be achieved indicating patients experiencing mild to moderate symptoms and functioning pretty well in daily life.
Adult patients : general functioning at 6 months | 6 months after randomization
  for Global assessment of functioning scale (GAF scale), a mean score of 60 and above is expected to be achieved indicating patients experiencing mild to moderate symptoms and functioning pretty well in daily life.
Adult patients : general functioning at 12 months | 12 months after randomization
  for Global assessment of functioning scale (GAF scale), a mean score of 60 and above is expected to be achieved indicating patients experiencing mild to moderate symptoms and functioning pretty well in daily life.
Minor patients : Child behaviour check list (CBCL) /6-18 scale at 1 month | 1 month after randomization
  For children>6 years old with an acute first episode or relapse of psychotic disorders: clinically significant difference ≤3 from baseline of CBCL/6-18 (Child Behavior Checklist) scale.
Minor patients : Child behaviour check list (CBCL) /6-18 scale at 3 months | 3 months after randomization
  For children>6 years old with an acute first episode or relapse of psychotic disorders: clinically significant difference ≤3 from baseline of CBCL/6-18 (Child Behavior Checklist) scale.
Minor patients : Child behaviour check list (CBCL) /6-18 scale at 6 months | 6 months after randomization
  For children>6 years old with an acute first episode or relapse of psychotic disorders: clinically significant difference ≤3 from baseline of CBCL/6-18 (Child Behavior Checklist) scale.
Minor patients : Child behaviour check list (CBCL) /6-18 scale at 12 months | 12 months after randomization
  For children>6 years old with an acute first episode or relapse of psychotic disorders: clinically significant difference ≤3 from baseline of CBCL/6-18 (Child Behavior Checklist) scale.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric VILLEGA, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (9):
- France (9):
  - Centre Hospitalier Charles Perrens, Bordeaux
  - CHU de Bordeaux, Bordeaux
  - Centre hospitalier le Vinatier, Bron
  - CHU de Clermond Ferrand, Clermont-Ferrand
  - APHP Louis Mourier, Colombes
  - APHP Henri Mondor, Créteil
  - APHP Kremlin Bicetre, Le Kremlin-Bicêtre
  - CHU de Montpellier, Montpellier
  - CHU de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No